CLINICAL TRIAL: NCT02849561
Title: Evaluation of Prognosis Factors of Neurological Evolution in Cardiac Arrest : Prospective Study of Routine Care
Brief Title: Evaluation of Prognosis Factors of Neurological Evolution in Cardiac Arrest
Acronym: ACR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 38RC13.713
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Cardio Respiratory Arrest
Keywords: Pupillary light reflex; Cardio respiratory arrest
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Favourable neurological evolution after cardiac arrest (Active Comparator): MGOS 4-5
  Interventions: Other: Therapeutic hypothermia; Device: Synchronized Intermittent Mandatory Ventilation; Other: Electroencephalography; Device: Pupillary light reflex surveillance; Device: Transcranial Doppler
- Unfavourable neurological evolution after cardiac arrest (Active Comparator): MGOS 1-3
  Interventions: Other: Therapeutic hypothermia; Device: Synchronized Intermittent Mandatory Ventilation; Other: Electroencephalography; Device: Pupillary light reflex surveillance; Device: Transcranial Doppler

INTERVENTIONS:
Other: Therapeutic hypothermia — With a mattress at 4°C to reach a central temperature at 33,5°C.
Device: Synchronized Intermittent Mandatory Ventilation — Constant volume 6 ml/kg
  Other Names: SIMV
Other: Electroencephalography
  Other Names: EEG
Device: Pupillary light reflex surveillance — With Neurolight® device.
Device: Transcranial Doppler — Monitoring tool for brain hemodynamic evaluation. With Philips HD15 Ultrasound system®.

SUMMARY:
With the repercussion of 55 cases eachyear for 100 000 inhabitants in France, cardio respiratory arrest is a public health issue.

The goal of this study is to evaluate the pupillary light reflex measured by the dimension of the pupil (diameter) as a prognosis factor neurological evolution in post cardiac arrest. By participating to this study, the patient get the same tratments and exams than in a usual managing cares.

In addition of these events, the pupillary light reflex is studied as soon as the patient is accepted in the department, and then on the second day.

Currently, the evaluation of the neurological becoming rely on a multimodal clinical and paraclinical approach.

The study of the pupillary light reflex measured by the diameter of the pupil could be a prognosis factor of neurological evolution for patients in post cardiac arrest, so a reliable and available prognosis marker in patient care.

The goal of this study is to evaluate the pupillary light reflex (RPM), measured by the diameter of the pupil as a prognosis factor of neurological evaluation of admitted patients after a cardiac arrest.

Principal criteria of judgement is the percentage of the pupillary light reflex variation measured with Neurolight®, compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Entry in resuscitation after a cardiac arrest intra or extra-hospital
* Resumption of a spontaneous cardiac activity
* Affiliation to a social security system

Exclusion Criteria:

* Refusal from patient or his family
* Age under 18 years
* Pregnant women
* Previous neurological damages
* Persons deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percentage of the pupillary light reflex variation measured with Neurolight® | One second
  Compared between two groups. Favourable neurological evolution after cardiac arrest : MGOS 4-5 Unfavourable neurological evolution after cardiac arrest MGOS 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Michel Durand, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Gorgels AP, Gijsbers C, de Vreede-Swagemakers J, Lousberg A, Wellens HJ. Out-of-hospital cardiac arrest--the relevance of heart failure. The Maastricht Circulatory Arrest Registry. Eur Heart J. 2003 Jul;24(13):1204-9. doi: 10.1016/s0195-668x(03)00191-x. PMID 12831814
- [Background] Jennett B, Plum F. Persistent vegetative state after brain damage. A syndrome in search of a name. Lancet. 1972 Apr 1;1(7753):734-7. doi: 10.1016/s0140-6736(72)90242-5. No abstract available. PMID 4111204
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Rogove HJ, Safar P, Sutton-Tyrrell K, Abramson NS. Old age does not negate good cerebral outcome after cardiopulmonary resuscitation: analyses from the brain resuscitation clinical trials. The Brain Resuscitation Clinical Trial I and II Study Groups. Crit Care Med. 1995 Jan;23(1):18-25. doi: 10.1097/00003246-199501000-00007. PMID 8001370
- [Background] Wijdicks EF, Hijdra A, Young GB, Bassetti CL, Wiebe S; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: prediction of outcome in comatose survivors after cardiopulmonary resuscitation (an evidence-based review) [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2006 Jul 25;67(2):203-10. doi: 10.1212/01.wnl.0000227183.21314.cd. PMID 16864809
- [Background] Edgren E, Hedstrand U, Kelsey S, Sutton-Tyrrell K, Safar P. Assessment of neurological prognosis in comatose survivors of cardiac arrest. BRCT I Study Group. Lancet. 1994 Apr 30;343(8905):1055-9. doi: 10.1016/s0140-6736(94)90179-1. PMID 7909098
- [Background] Kamps MJ, Horn J, Oddo M, Fugate JE, Storm C, Cronberg T, Wijman CA, Wu O, Binnekade JM, Hoedemaekers CW. Prognostication of neurologic outcome in cardiac arrest patients after mild therapeutic hypothermia: a meta-analysis of the current literature. Intensive Care Med. 2013 Oct;39(10):1671-82. doi: 10.1007/s00134-013-3004-y. Epub 2013 Jun 26. PMID 23801384
- [Background] Fischer C, Luaute J, Nemoz C, Morlet D, Kirkorian G, Mauguiere F. Improved prediction of awakening or nonawakening from severe anoxic coma using tree-based classification analysis. Crit Care Med. 2006 May;34(5):1520-4. doi: 10.1097/01.CCM.0000215823.36344.99. PMID 16557163
- [Background] Jorgensen EO. Course of neurological recovery and cerebral prognostic signs during cardio-pulmonary resuscitation. Resuscitation. 1997 Aug;35(1):9-16. doi: 10.1016/s0300-9572(97)00022-1. PMID 9259054
- [Background] Meeker M, Du R, Bacchetti P, Privitera CM, Larson MD, Holland MC, Manley G. Pupil examination: validity and clinical utility of an automated pupillometer. J Neurosci Nurs. 2005 Feb;37(1):34-40. PMID 15794443
- [Background] Behrends M, Niemann CU, Larson MD. Infrared pupillometry to detect the light reflex during cardiopulmonary resuscitation: a case series. Resuscitation. 2012 Oct;83(10):1223-8. doi: 10.1016/j.resuscitation.2012.05.013. Epub 2012 May 30. PMID 22659054
- [Background] Taylor WR, Chen JW, Meltzer H, Gennarelli TA, Kelbch C, Knowlton S, Richardson J, Lutch MJ, Farin A, Hults KN, Marshall LF. Quantitative pupillometry, a new technology: normative data and preliminary observations in patients with acute head injury. Technical note. J Neurosurg. 2003 Jan;98(1):205-13. doi: 10.3171/jns.2003.98.1.0205. PMID 12546375
- [Background] Horburger D, Testori C, Sterz F, Herkner H, Krizanac D, Uray T, Schober A, Stockl M, Stratil P, Weiser C, Wallmuller C, Holzer M. Mild therapeutic hypothermia improves outcomes compared with normothermia in cardiac-arrest patients--a retrospective chart review. Crit Care Med. 2012 Aug;40(8):2315-9. doi: 10.1097/CCM.0b013e31825333cf. PMID 22622403
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Nunnally ME, Jaeschke R, Bellingan GJ, Lacroix J, Mourvillier B, Rodriguez-Vega GM, Rubertsson S, Vassilakopoulos T, Weinert C, Zanotti-Cavazzoni S, Buchman TG. Targeted temperature management in critical care: a report and recommendations from five professional societies. Crit Care Med. 2011 May;39(5):1113-25. doi: 10.1097/CCM.0b013e318206bab2. PMID 21187745
- [Background] Nolan JP, Neumar RW, Adrie C, Aibiki M, Berg RA, Bbttiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T; International Liaison Committee on Resuscitation; Emergency Cardiovascular Care Committee, American Heart Association; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiopulmonary, Perioperative, and Critical Care; Council on Clinical Cardiology; Council on Stroke. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication: a scientific statement from the International Liaison Committee on Resuscitation; the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; the Council on Stroke (Part II). Int Emerg Nurs. 2010 Jan;18(1):8-28. doi: 10.1016/j.ienj.2009.07.001. Epub 2009 Aug 5. PMID 20129438
- [Background] Gueugniaud PY, Garcia-Darennes F, Gaussorgues P, Bancalari G, Petit P, Robert D. Prognostic significance of early intracranial and cerebral perfusion pressures in post-cardiac arrest anoxic coma. Intensive Care Med. 1991;17(7):392-8. doi: 10.1007/BF01720676. PMID 1774392
- [Background] Alvarez-Fernandez JA. [Transcranial Doppler ultrasound use in post-cardiac arrest coma]. Rev Neurol. 2011 Nov 1;53(9):545-54. Spanish. PMID 22012818
- [Background] Wessels T, Harrer JU, Jacke C, Janssens U, Klotzsch C. The prognostic value of early transcranial Doppler ultrasound following cardiopulmonary resuscitation. Ultrasound Med Biol. 2006 Dec;32(12):1845-51. doi: 10.1016/j.ultrasmedbio.2006.06.023. PMID 17169697
- [Background] Edgren E, Hedstrand U, Nordin M, Rydin E, Ronquist G. Prediction of outcome after cardiac arrest. Crit Care Med. 1987 Sep;15(9):820-5. doi: 10.1097/00003246-198709000-00004. PMID 3621954
- [Background] Zandbergen EG, de Haan RJ, Stoutenbeek CP, Koelman JH, Hijdra A. Systematic review of early prediction of poor outcome in anoxic-ischaemic coma. Lancet. 1998 Dec 5;352(9143):1808-12. doi: 10.1016/S0140-6736(98)04076-8. PMID 9851380
- [Background] Zandbergen EG, Koelman JH, de Haan RJ, Hijdra A; PROPAC-Study Group. SSEPs and prognosis in postanoxic coma: only short or also long latency responses? Neurology. 2006 Aug 22;67(4):583-6. doi: 10.1212/01.wnl.0000230162.35249.7f. PMID 16924008
- [Background] Nakabayashi M, Kurokawa A, Yamamoto Y. Immediate prediction of recovery of consciousness after cardiac arrest. Intensive Care Med. 2001 Jul;27(7):1210-4. doi: 10.1007/s001340100984. PMID 11534570
- [Background] Rothstein TL. The role of evoked potentials in anoxic-ischemic coma and severe brain trauma. J Clin Neurophysiol. 2000 Sep;17(5):486-97. doi: 10.1097/00004691-200009000-00007. PMID 11085552
- [Background] Vanhaudenhuyse A, Laureys S, Perrin F. Cognitive event-related potentials in comatose and post-comatose states. Neurocrit Care. 2008;8(2):262-70. doi: 10.1007/s12028-007-9016-0. PMID 17990124
- [Background] Tzovara A, Rossetti AO, Spierer L, Grivel J, Murray MM, Oddo M, De Lucia M. Progression of auditory discrimination based on neural decoding predicts awakening from coma. Brain. 2013 Jan;136(Pt 1):81-9. doi: 10.1093/brain/aws264. Epub 2012 Nov 12. PMID 23148350
- [Background] Cummins RO, Chamberlain DA, Abramson NS, Allen M, Baskett PJ, Becker L, Bossaert L, Delooz HH, Dick WF, Eisenberg MS, et al. Recommended guidelines for uniform reporting of data from out-of-hospital cardiac arrest: the Utstein Style. A statement for health professionals from a task force of the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, and the Australian Resuscitation Council. Circulation. 1991 Aug;84(2):960-75. doi: 10.1161/01.cir.84.2.960. No abstract available. PMID 1860248
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Rana OR, Schroder JW, Kuhnen JS, Saygili E, Gemein C, Zink MD, Schauerte P, Schiefer J, Schwinger RH, Weis J, Marx N, Kelm M, Meyer C, Saygili E. The Modified Glasgow Outcome Score for the prediction of outcome in patients after cardiac arrest: a prospective clinical proof of concept study. Clin Res Cardiol. 2012 Jul;101(7):533-43. doi: 10.1007/s00392-012-0423-7. Epub 2012 Feb 10. PMID 22322567
- [Background] Bouzat P, Suys T, Sala N, Oddo M. Effect of moderate hyperventilation and induced hypertension on cerebral tissue oxygenation after cardiac arrest and therapeutic hypothermia. Resuscitation. 2013 Nov;84(11):1540-5. doi: 10.1016/j.resuscitation.2013.05.014. Epub 2013 May 30. PMID 23727361